CLINICAL TRIAL: NCT03949348
Title: Transobturator Urethral Sling Placement With an Autologous Rectus Facia for Female Stress Urinary Incontinence.
Brief Title: Transobturator Urethral Sling Placement With an Autologous Rectus Facia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal invastigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0635
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Stress Urinary Incontinence; Surgery--Complications
Keywords: midurethral sling placement; synthetic mesh; autologous rectus fascia; transobturator approach
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Patients who undergo a transobturator sling placement using autologous rectus fascia
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous fascia (Active Comparator): Patients who underwent a transobturator sling placement using autologous rectus fascia
  Interventions: Procedure: Mid-urethral sling placement using autologous rectus fascia
- synthetic mesh (Active Comparator): Patients who underwent a transobturator sling placement using synthetic mesh
  Interventions: Procedure: Mid-urethral sling placement using synthetic mesh

INTERVENTIONS:
Procedure: Mid-urethral sling placement using autologous rectus fascia — Mid-urethral sling placement using autologous rectus fascia
  Arms: autologous fascia
Procedure: Mid-urethral sling placement using synthetic mesh — Mid-urethral sling placement using synthetic mesh
  Arms: synthetic mesh

SUMMARY:
The investigators aimed to evaluate outcomes of transobturator urethral sling placement using autologous rectus fascia for female stress urinary incontinence at perioperatively and at 2-year follow-up.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is very common condition in middle-aged women, and can affect quality of life. Some clinical trials reported that the lifetime risk of a woman undergoing surgery for SUI is increase in up to 15%. The midurethral synthetic sling is the most common surgery performed for female SUI. This procedure has high efficacy and low perioperative morbidity.

Although many clinical trials have demonstrated that synthetic mid-urethral slings are safe, effective and recommended by several guidelines (e.g. Society of Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction/American Urogynecologic Society and American Urologic Association), the safety and efficacy of surgery for SUI using mesh devices has been questioned by a community of patients and clinicians. After Food and Drug Administration notification on mesh use in pelvic surgery, many patients and providers begin to search of different surgery without synthetic mesh alternatives in SUI. Recently, female patients in England formed the campaign group "Sling the Mesh" to protest the synthetic mesh.

Several options such as the autologous pubovaginal sling, biologic grafts, or urethral bulking agent injection have some problems related to morbidity or efficacy. The autologous pubovaginal urethral sling is associated with a higher risk of postoperative voiding dysfunction.

The investigators aimed to demonstrate the feasibility of an autologous transobturator urethral sling to avoid the related problems of synthetic mesh placement and the increased rate of voiding dysfunction with pubovaginal sling placement.

ELIGIBILITY:
Inclusion Criteria:

* female patients that underwent mid-urethral sling placement

Exclusion Criteria:

* active urinary infection
* neurologic disorders
* malignancies
* history of radiotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Surgery for female stress urinary incontinence
Enrollment: 35 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
ICIQ-SF | 2 years
  The ICIQ-UI Short Form is a brief and psychometrically robust patient-completed questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in women in research and clinical practice across the world. It is scored on a scale from 0-21; higher values represent worse outcomes. The ICIQ-UI Short Form provides a brief and robust measure to assess the impact of symptoms of incontinence on outcome.

SECONDARY OUTCOMES:
Treatment Benefit Scale | 2 years
  TBS consists of four categories scored as 1 (greatly improved) or 2 (improved), considered as ''yes,'' or 3 (not changed) or 4 (worsened), which were considered as ''no''

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Linder BJ, Elliott DS. Autologous Transobturator Urethral Sling Placement for Female Stress Urinary Incontinence: Short-term Outcomes. Urology. 2016 Jul;93:55-9. doi: 10.1016/j.urology.2016.03.025. Epub 2016 Mar 29. PMID 27036519
- [Result] Linder BJ, Elliott DS. Autologous transobturator urethral sling placement for female stress urinary incontinence. J Urol. 2015 Mar;193(3):991-6. doi: 10.1016/j.juro.2014.08.125. Epub 2014 Oct 19. PMID 25444955